CLINICAL TRIAL: NCT05699057
Title: Prevalence and Associated Risk Factors of Tendency to Suicide as a Sequel of Computer Vision Syndrome Among Medical Students in Egypt
Brief Title: Tendency to Suicide as a Sequel of Computer Vision Syndrome
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Professor of Ophthalmology, Sohag University
Other Study IDs: Soh-Med-22-10-25
Record Dates: First submitted 2022-10-09; First posted 2023-01-26 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Suicide GROUP — CVS-F4 will be an online survey via the SurveyMonkey Company. The participants will report their potential CVS complains and associated screen factors as screen-time, screen-size, screen-resolution and other factors. We will collect the responses and analyse the results. Informed consent will be obtained from the participants as an item within the survey itself that he/she agrees to use his/her data in this research work. This group will contain participants with CVS complains. Finally, we will To document the prevalence of tendency to suicide among medical students in the Egyptian Universities and analyse associated risk factors and any correlated determents.

SUMMARY:
CVS-F4 questionnaire will be used as an instrument to survey prevalence of tendency to suicide among medical students in the Egyptian Universities and analyse associated risk factors and any correlated determents

DETAILED DESCRIPTION:
CVS-F4 (30 questions) will be an online survey via the SurveyMonkey Company. We will collect the responses and analyze the results. Informed consent will be obtained from the participants as an item within the survey itself that he/she agrees to use his/her data in this research work. The questionnaire includes questions regarding potential ocular, extra-ocular, musclo-skeletal and neuro-psychatric complains caused by CVS. CVS-F4 questionnaire will be used as an instrument to survey prevalence of tendency to suicide among medical students in the Egyptian Universities and analyse associated risk factors and any correlated determents Complete statistical analysis of the survey data will be done using univariate and multivariate logistic and linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* university students
* university staff members

Exclusion Criteria:

* hysteria
* ocular surgery
* amblyopia
* anisometropia
* strabismus
* systemic disease

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: medical students or staff who are using screens in their medical studies or personal lives and how these screens affect their medical studies and the effect of mandated medical computer use if present on their screen-behaviour, tendency to suicide and associated risk factor
Sampling Method: Probability Sample
Enrollment: 3512 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Tendency to suicide | 3 months
  The participants will respond to Computer Vision Syndrome (CVS-F4) questionnaire and the number and percentage of participants suffering from tendency to suicide will be recorded
Depression | 3 months
  The participants will respond to Computer Vision Syndrome (CVS-F4) questionnaire and the number and percentages of participants suffering from tendency to suicide and depression will be recorded. A correlation between depression and tendency to suicide will be measured as P value less than 0.05 will be significant
Screen-time | 3 months
  The total daily average screen-hours will be measured using mean and standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal Iqbal, MD, PhD, Principal Investigator — Professor of Ophthalmology
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study data will available at the principal investigator for other researchers upon reasonable request after publication of the study
Supporting Information: Study Protocol, CSR
Time Frame: 12 months